CLINICAL TRIAL: NCT04098276
Title: An Adaptive Intervention to Improve Health, Safety and Empowerment Outcomes Among Immigrant Women With Intimate Partner Violence Experiences
Brief Title: It's WeWomen Plus Intervention for Health, Safety and Empowerment
Acronym: IWWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00224324; R01MD013863-01A1 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Violence, Domestic; Violence-Related Symptom; Violence, Physical; Violence, Sexual; Violence, Gender-Based; Violence
Keywords: Intimate partner violence; safety planning; immigrant; risk for future violence; risk for intimate partner homicide; empowerment; mental health; safety
MeSH Terms: conditions — Coitus; Empowerment; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study used a sequential, multiple assignment, randomized (SMART) design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Personalized Online Intervention (Experimental): For first stage randomization, women in the personalized online intervention group receive the online safety planning intervention informed by culturally specific danger assessment (DA) tool.
  Interventions: Behavioral: WeWomen Plus technology based intervention
- Online usual care or Standard Online Safety Information (No Intervention): Women in the Standard Online Safety Information received the non-DA informed usual safety planning resources modeled on national and state domestic violence online resources, but not provided with immediate and visual feedback to their level of danger or a tailored safety planning.
- WeWomen Plus Text messaging only (Experimental): For second stage randomization, the text messaging intervention will follow-up with non-responder group of immigrant women (those who did not improve in intervention or control arms above) on their enactment of tailored (tailored to the DA Score and priorities) safety plan provided in the online weWomen intervention or non-tailored (standard list of resources) safety recommendations provided in the usual care control arm
  Interventions: Behavioral: WeWomen Plus technology based intervention
- WeWomen Plus Text messaging and phone (Experimental): Second stage randomization will involve both text (described above) and phone calls for non-responder group of women in intervention or control arm. The phone calls will draw from motivational interviewing adapted for abused women, solution focused therapy and a strengths perspective to discuss women's safety concerns and other needs, and strategies to strengthen social support networks
  Interventions: Behavioral: WeWomen Plus technology based intervention

INTERVENTIONS:
Behavioral: WeWomen Plus technology based intervention — The WeWomen Plus intervention is a technology based (online, text and phone)culturally tailored intervention designed to reduce the risk of future intimate partner violence or a homicide, improve mental health and increase empowerment of abused immigrant women.
  Arms: Personalized Online Intervention; WeWomen Plus Text messaging and phone; WeWomen Plus Text messaging only

SUMMARY:
This study evaluates the impact of adaptive technology-based intervention (online, text and phone) "weWomenPlus" on safety, mental health and empowerment of abused immigrant women.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) disproportionately affects immigrant women. However, immigrant women remain an understudied and underserved population in need for evidence-based rigorously evaluated culturally competent interventions that address the health and safety needs of immigrant women. This study used a sequential, multiple assignment, randomized trial (SMART) design to rigorously evaluate an adaptive culturally informed intervention tailored to needs of immigrant women with IPV experiences. For the first stage randomization, participants were randomly assigned to a personalized online intervention or the standard online safety information/usual care control arm and safety, mental health and empowerment outcomes were assessed at 3, 6 and 12 months follow up. For the second stage randomization, women who did not report significant improvement in safety (i.e., reduction in IPV) and in empowerment from baseline to follow up points (i.e., non-responders) were re- randomized to the augmented intervention components (text only or a combination of text and phone) developed in the formative phase. Data on outcomes (safety, mental health and empowerment) were assessed at 6 and 12 months of re- randomization. By re-randomizing participants, the study assessed the relative effectiveness of two strategies for augmentation (text only or a combination of text and phone) on safety, mental health and empowerment outcomes among the non-responders of the online interventions. In addition, the study compared the non-responder group of women to the responder group of the online interventions to determine if the strategies of augmentation brought the non-responders to the level of responders on safety, mental health and empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Experiences of intimate partner violence within the past one year
* Foreign born immigrant woman
* 18-64 years of age
* Can access and use internet and phone

Exclusion Criteria:

* No experience of intimate partner violence within the past one year
* US born
* Younger than 18 or older than 64
* Cannot access or use internet or phone

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 1265 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sabri, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Sabri B, Glass N, Murray S, Perrin N, Case JR, Campbell JC. A technology-based intervention to improve safety, mental health and empowerment outcomes for immigrant women with intimate partner violence experiences: it's weWomen plus sequential multiple assignment randomized trial (SMART) protocol. BMC Public Health. 2021 Oct 28;21(1):1956. doi: 10.1186/s12889-021-11930-2. PMID 34711182
- Available data/document: Study Protocol: 10.1186/s12889-021-11930-2 — https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-021-11930-2

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Online Intervention: For first stage randomization, women in the personalized online intervention group receive the online safety planning intervention informed by culturally specific danger assessment (DA) tool.
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology-based (online, text, and phone) intervention designed to reduce the risk of future intimate partner violence or homicide, improve mental health, and increase the empowerment of abused women.
- Online Usual Care or Standard Online Safety Information: Women in the Standard Online Safety Information condition received the non-DA informed usual safety planning resources modeled on national and state domestic violence online resources but not provided with immediate and visual feedback to their level of danger or a tailored safety planning.
- WeWomen Plus Text Messaging Only: For second stage randomization, the text messaging intervention followed-up with non-responder group of immigrant women (those who did not improve in intervention or control arms above) on their enactment of tailored (tailored to the DA Score and priorities) safety plan provided in the personalized online intervention or non-tailored (standard list of resources) safety recommendations provided in the usual care or standard online safety information arm.
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology-based (online, text, and phone) intervention designed to reduce the risk of future intimate partner violence or homicide, improve mental health, and increase empowerment of abused women.
- WeWomen Plus Text Messaging and Phone: Second-stage randomization involved both text and phone calls for non-responder groups of women in personalized online or standard online safety information arm. The phone calls will draw from motivational interviewing adapted for abused women, solution-focused therapy, and a strengths perspective to discuss women's safety concerns and other needs and strategies to strengthen social support networks
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology-based (online, text, and phone) intervention designed to reduce the risk of future intimate partner violence or homicide, improve mental health, and increase empowerment of abused women.
Period: First Stage Randomization
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Started | 660 | 605 | 0 | 0
Completed | 618 | 573 | 0 | 0
Not Completed | 42 | 32 | 0 | 0
Period: Second Stage Re-Randomization
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Started (Women who did not show significant improvement in the first-stage intervention were re-randomized to second-stage interventions. Specifically, 183 unique participants were re-randomized to WeWomen Plus Text Messaging Only arm and a different 183 unique participants were re-randomized to WeWomen Plus Text Messaging and Phone arm (366 total re-randomized participants).) | 0 | 0 | 183 | 183
Completed | 0 | 0 | 165 | 156
Not Completed | 0 | 0 | 18 | 27

BASELINE CHARACTERISTICS:
Groups:
- Personalized Online Intervention: Women received the culturally adapted myPlan intervention, a web-based safety decision-making tool based on Dutton's empowerment model with danger assessment and tailored safety planning.
- Standard Online Safety Information: Women received usual safety planning resources modeled on national and state domestic violence online resources without danger assessment-informed safety planning.
- Total: Total of all reporting groups
Arm/Group | Personalized Online Intervention | Standard Online Safety Information | Total
Number analyzed (Participants) | 660 | 605 | 1265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 14
  Between 18 and 65 years | 652 | 599 | 1251
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.70 (9.88) | 37.39 (9.67) | 37.00 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 660 | 605 | 1265
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 255 | 269 | 524
  Not Hispanic or Latino | 396 | 330 | 726
  Unknown or Not Reported | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 222 | 164 | 386
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 85 | 87 | 172
  White | 167 | 189 | 356
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 181 | 159 | 340
Physical and Sexual IPV [Mean (Standard Deviation); unit: units on a scale] — Physical and sexual intimate partner violence (IPV) was measured using the adapted version of the Revised Conflict Tactics Scale (CTS2), with response categories ranging from 0=never to 4=very frequently. Total score ranged from 0-164, with higher scores indicating greater frequency and severity of intimate partner violence experiences.
  units on a scale | 18.03 (25.52) | 17.83 (25.07) | 17.94 (25.29)
Depression [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms were measured using The Patient Health Questionnaire (PHQ-9), a nine-item measure. Each of the nine items scored from 0 (not at all) to 3 (nearly every day). Total scores ranged from 0 to 27, with higher scores indicating more severe depression symptoms. A score of 10 or above indicates clinically significant depression symptoms.
  units on a scale | 9.98 (6.39) | 10.39 (6.61) | 10.18 (6.50)
Post-traumatic Stress Disorder (PTSD) [Mean (Standard Deviation); unit: units on a scale] — Past week PTSD symptoms were measured using the Harvard Trauma Questionnaire (16 items), with response options ranging from 1 (Not at all) to 5 (Extremely) per item. The mean of the participant scale choices (1-5) across all 16 items is reported. Higher scores indicated more severe PTSD symptoms, with score greater than 2.5 indicating clinically significant PTSD symptoms.
  units on a scale | 2.42 (0.93) | 2.50 (1) | 2.46 (0.96)
Overall Empowerment [Mean (Standard Deviation); unit: units on a scale] — The Personal Progress Scale-Revised (PPS-R) (23 items) was used to assess multiple areas associated with overall empowerment. The responses were rated on a 7-point scale ranging from 1 (almost Never) to 7 (almost Always). The scores ranged from 23 to 161. Higher scores indicated a higher level of empowerment.
  units on a scale | 119.60 (21.19) | 118.85 (21.67) | 119.24 (21.41)
Safety-Related Empowerment [Mean (Standard Deviation); unit: units on a scale] — The MOVERS, a 13-item scale, was used to measure empowerment within the domain of safety. Participants responded to each item using a five-point scale, ranging from "1 = never true" to "5 = always true". The mean of the participant scale choices (1-5) across all 13 items is reported. Higher scores indicated a greater degree of safety-related empowerment.
  units on a scale | 3.36 (0.72) | 3.38 (0.75) | 3.37 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Physical and Sexual Intimate Partner Violence as Assessed by the Revised Conflict Tactics Scale
Description: The adapted version of the Revised Conflict Tactics Scale (CTS2; Straus, 1996) was used to measure the severity and frequency of abusive or violent acts in intimate partner relationships. The CTS2 subscales included physical aggression, injury, psychological aggression, and sexual coercion. Response categories ranged from 0=never to 4=very frequently. Total scores ranged from 0-164, with higher scores indicating greater frequency and severity of intimate partner violence experiences. Items were scored using the severity-times-frequency weighted score method as recommended by Straus (1996). Change scores were calculated as the differences between baseline CTS-2 total scores and follow-up scores at each time point (3, 6, and 12 months).
Time Frame: Baseline (1st month), 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Personalized Online Intervention: For first stage randomization, women in the personalized online intervention group receive the online safety planning intervention informed by culturally specific danger assessment (DA) tool.
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology based (online, text and phone) culturally tailored intervention designed to reduce the risk of future intimate partner violence or a homicide, improve mental health and increase empowerment of abused immigrant women.
- Online Usual Care or Standard Online Safety Information: Women in the Standard Online Safety Information received the non-DA informed usual safety planning resources modeled on national and state domestic violence online resources but not provided with immediate and visual feedback to their level of danger or a tailored safety planning.
- WeWomen Plus Text Messaging Only: For second stage randomization, the text messaging intervention will follow-up with non-responder group of immigrant women (those who did not improve in intervention or control arms above) on their enactment of tailored (tailored to the DA Score and priorities) safety plan provided in the online weWomen intervention, or non-tailored (standard list of resources) safety recommendations provided in the usual care control arm
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology based (online, text and phone) culturally tailored intervention designed to reduce the risk of future intimate partner violence or a homicide, improve mental health and increase empowerment of abused immigrant women.
- WeWomen Plus Text Messaging and Phone: Second stage randomization will involve both text (described above) and phone calls for non-responder group of women in intervention or control arm. The phone calls will draw from motivational interviewing adapted for abused women, solution focused therapy and a strengths perspective to discuss women's safety concerns and other needs, and strategies to strengthen social support networks
  WeWomen Plus technology-based intervention: The WeWomen Plus intervention is a technology based (online, text and phone) culturally tailored intervention designed to reduce the risk of future intimate partner violence or a homicide, improve mental health and increase empowerment of abused immigrant women.
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Number analyzed (Participants) | 660 | 605 | 183 | 183
score on a scale
  1-3 months | -6.29 (22.56) | -5.16 (21.07) | -2.20 (20.01) | -1.82 (21.30)
  1-6 months | -7.65 (22.35) | -5.62 (21.61) | -4.61 (20.63) | -8.27 (20.87)
  3- 6 months | -0.81 (16.07) | -0.30 (18.96) | -1.74 (20.99) | -6.10 (19.33)
  3 -12 months | -0.24 (20.81) | 0.03 (19.47) | -0.43 (19.73) | -4.94 (24.50)
  1-12 months | -6.46 (22.15) | -5.22 (22.50) | -3.50 (23.34) | -7.27 (22.32)

2. Secondary Outcome: Change in Depressive Symptoms as Assessed by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) was used to assess depression symptoms over the past two weeks based on DSM-IV diagnostic criteria for major depressive disorder. Each of the 9 items was scored from 0 (not at all) to 3 (nearly every day). Total scores were computed by summing all items, ranging from 0-27. Higher scores indicated more severe depression symptoms (1-4=minimal, 5-9=mild, 10-14=moderate, 15-19=moderately severe, 20-27=severe depression). Change scores were calculated as the differences between baseline PHQ-9 total scores and follow-up scores at each time point (3, 6, and 12 months).
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Number analyzed (Participants) | 660 | 605 | 183 | 183
score on a scale
  1-3 months | -0.41 (5.32) | -0.35 (5.23) | 0.83 (5.35) | 0.03 (4.71)
  1-6 months | -1.04 (5.61) | -1.45 (5.79) | -1.20 (5.90) | -1.41 (5.58)
  3-6 months | -0.66 (5.36) | -1.07 (5.43) | -2.02 (5.47) | -1.51 (5.41)
  3-12 months | -0.87 (5.97) | -0.87 (5.66) | -1.79 (5.88) | -1.78 (5.70)
  1-12 months | -1.20 (6.18) | -1.25 (6.02) | -0.95 (5.82) | -1.73 (5.31)

3. Secondary Outcome: Change in Symptoms of Post-traumatic Stress Disorder (PTSD) as Assessed by the Harvard Trauma Questionnaire
Description: Past week PTSD symptoms were measured using the Harvard Trauma Questionnaire, a 16-item scale with response options that ranged from 1 (not at all) to 5 (extremely). Mean scores across all 16 items were calculated for each participant. Higher scores indicated more severe PTSD symptoms, with scores greater than 2.5 indicating clinically significant PTSD symptoms. Change scores were calculated as the differences between baseline mean scores and the follow-up mean scores at each time point (3, 6, and 12 months).
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Number analyzed (Participants) | 660 | 605 | 183 | 183
score on a scale
  1-3 months | -0.10 (0.75) | -0.11 (0.76) | 0.01 (0.76) | -0.09 (0.73)
  3-6 months | -0.08 (0.71) | -0.06 (0.72) | -0.22 (0.79) | -0.09 (0.79)
  1-6 months | -0.18 (0.78) | -0.18 (0.78) | -0.24 (0.87) | -0.19 (0.74)
  3-12 months | -0.08 (0.81) | -0.04 (0.76) | -0.18 (0.83) | -0.14 (0.81)
  1-12 months | -0.18 (0.82) | -0.17 (0.88) | -0.16 (0.82) | -0.27 (0.87)

4. Secondary Outcome: Change in Overall Empowerment as Assessed by the Personal Progress Scale-Revised
Description: The Personal Progress Scale-Revised was used to measure empowerment across multiple domains including positive self-evaluation, self-esteem, emotional regulation, gender-role and cultural identity awareness, self-efficacy, self-care, problem-solving, and assertiveness skills. Participants rated 28 items on a 7-point scale from 1 (almost never) to 7 (almost always). Total scores were calculated by summing all items, ranging from 28-196, with higher scores indicating greater empowerment. Change scores were calculated as the differences between baseline total scores and follow-up scores at each time point (3, 6, and 12 months).
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Number analyzed (Participants) | 660 | 605 | 183 | 183
score on a scale
  1-3 months | 0.42 (16.30) | 0.66 (16.76) | -3.16 (15.89) | -5.10 (15.92)
  3-6 months | 1.20 (16.01) | 1.20 (15.73) | 2.74 (16.20) | 5.35 (16.71)
  1-6 months | 1.20 (17.81) | 1.81 (17.41) | -0.39 (16.23) | -0.05 (16.63)
  3-12 months | 1.46 (17.80) | -0.53 (16.62) | 2.59 (15.47) | 3.75 (16.85)
  1-12 months | 1.25 (20.52) | 0.33 (18.25) | -0.84 (17.09) | -1.35 (17.66)

5. Secondary Outcome: Change in Empowerment Related to Safety as Assessed by the Measure of Victim Empowerment Related to Safety (MOVERS) Scale
Description: The MOVERS scale was used to measure empowerment within the safety domain, including safety-related goal development, self-efficacy beliefs, and knowledge of support resources. Participants rated 13 items on a 5-point scale from 1 (never true) to 5 (always true). Mean scores across all 13 items were calculated for each participant. Higher scores indicated greater safety-related empowerment. Change scores were calculated as the differences between baseline mean scores and follow-up mean scores at each time point (3, 6, and 12 months).
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
Number analyzed (Participants) | 660 | 605 | 183 | 183
score on a scale
  1-3 months | 0.16 (0.71) | 0.10 (0.69) | -0.40 (0.45) | -0.39 (0.45)
  3-6 months | -0.10 (0.70) | -0.06 (0.72) | 0.35 (0.64) | 0.29 (0.64)
  1-6 months | 0.08 (0.63) | 0.04 (0.65) | -0.04 (0.61) | -0.10 (0.63)
  3-12 months | -0.09 (0.70) | -0.09 (0.72) | 0.34 (0.63) | 0.24 (0.58)
  1-12 months | 0.07 (0.68) | 0.02 (0.71) | -0.07 (0.54) | -0.16 (0.66)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Personalized Online Intervention | Online Usual Care or Standard Online Safety Information | WeWomen Plus Text Messaging Only | WeWomen Plus Text Messaging and Phone
All-Cause Mortality (participants affected / at risk) | 0/660 | 0/605 | 0/183 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/660 | 0/605 | 0/183 | 0/183
Other Adverse Events (participants affected / at risk) | 0/660 | 0/605 | 0/183 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04098276/Prot_SAP_000.pdf